CLINICAL TRIAL: NCT01041430
Title: Randomized Clinical Trial Comparing Day-case and Inpatient Care Following Inguinal Hernia Repair in Elderly Patients
Brief Title: Day-case or Inpatient Care Following Inguinal Hernia Repair in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kristiina Mattila, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T102010087a
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Hernia, Inguinal
Keywords: Ambulatory Surgery; Aged
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day Surgery Group (Active Comparator): discharge planned on day of surgery, inguinal hernia repair
  Interventions: Other: day surgery group
- Inpatient Group (Active Comparator): overnight admission at the hospital, inguinal hernia repair
  Interventions: Other: inpatient group

INTERVENTIONS:
Other: day surgery group — inguinal hernia repair, discharge from the hospital on the day of surgery
  Arms: Day Surgery Group
Other: inpatient group — inguinal hernia repair, patient admitted overnight to hospital
  Arms: Inpatient Group

SUMMARY:
The aim of the study was to evaluate the feasibility of day surgery for elderly patients undergoing elective open inguinal hernia repair. Medically stable patients aged 65 years or older, with postoperative care available at home, were randomized to receive treatment either as day-cases or inpatients. Younger day-case patients undergoing the same procedure served as controls. Outcome measures during two postoperative weeks were complications, unplanned admissions and visits to the hospital, unplanned visits to primary health care and patients' acceptance of the type of provided care. The investigators expected to find a higher degree of satisfaction in the patient group receiving day-case care.

DETAILED DESCRIPTION:
For repair of inguinal hernia, standard open mesh repair methods were used. For anaesthesia, local infiltration with lidocaine (10 mg/ml) and light intravenous sedation with propofol and fentanyl were primarily used. Reasons for choosing spinal or general anaesthesia were registered. For postoperative pain relief bupivacaine (5mg/ml) 10 ml was infiltered into the wound and nonsteroidal anti-inflammatory analgesics (NSAID) and paracetamol combined with codeine were prescribed, when suitable. Day-case patients were discharged home according to commonly approved criteria. Inpatients stayed on the hospital ward overnight. All patients received the same preoperative and postoperative instructions orally and in writing. Physical activity was not restricted after the operation, and patients were encouraged to resume to normal life as soon as possible.

At the hospital, patient characteristics, type of anaesthesia, duration of surgery, duration of hospital stay and perioperative complications including unplanned overnight admissions were registered.

The study nurse interviewed all patients on the 1st and 14th postoperative day (POD) by telephone, using standardised follow-up questionnaires. The investigated variables on both dates included: satisfaction with treatment, patient-reported overall condition and functional capacity compared to the preoperative state, intensity of pain and use of pain medication. On POD 1, patients were inquired whether convalescence had been as expected, and asked to specify if not. Also the incidence and intensity other symptoms apart from pain were questioned. On POD 14 patients were questioned of unplanned contacts with primary healthcare, unplanned hospital visits, readmissions, and corresponding reasons.

Patient satisfaction with treatment in the operating room and following arrival to the postanaesthesia care unit was evaluated numerically (0-10), using the numeric rating scale (NRS), with 0 indicating lowest, and 10 highest possible satisfaction as rated by the patient. Intensity of postoperative pain was evaluated by NRS. Overall condition and functional capacity were evaluated using a 3 -point scale (good / moderate / poor). Health-related quality of life was measured using the RAND-36-instrument.

Patients were inquired about the degree of impairment in the groin area at the preoperative visit, and three months postoperatively.

Results are given as median (range) or mean (SD) as appropriate. Patient characteristics and surgery -related variables and NRS scores were compared using the Chi-square, Mann-Whitney-U and Kruskall-Wallis tests when appropriate. Intergroup comparisons were performed using the Wilcoxon test for related samples. P-values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* referral for open repair of inguinal hernia

Exclusion Criteria:

* severe comorbidity (ASA class IV, unstable ASA class III)
* postoperative care at home not available
* not willing to receive day-case care
* unable to understand numeric rating scale

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 2 weeks postoperatively
  satisfaction based on type of care

SECONDARY OUTCOMES:
short term outcome | 2 weeks postoperatively
  rate of complications, unplanned admissions, unplanned visits to the hospital, unplanned visits to primary health care

CONTACTS AND LOCATIONS:
Overall Officials: Kristiina Mattila, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Jorvi Hospital, Helsinki University Hospital, Espoo, HUS, Finland